CLINICAL TRIAL: NCT05090930
Title: Development of Innovative Technologies for the Treatment of Pulmonary and Heart Failure to Prolong Human's Life
Brief Title: Innovative Technologies for the Treatment of Pulmonary and Heart Failure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Research Center for Cardiac Surgery, Kazakhstan (Other)
Collaborators: Ministry of Education and Science, Republic of Kazakhstan (Other Government)
Responsible Party: Principal Investigator, Yuriy Pya, Director for Surgery and Science, National Research Center for Cardiac Surgery, Kazakhstan
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: version01; BR10965200 (Other Grant/Funding Number: Ministry of Education and Science RK)
Record Dates: First submitted 2021-09-09; First posted 2021-10-25 (Actual); Last update posted 2021-10-25 (Actual); Status verified 2021-10

CONDITIONS: Cardiogenic Shock; Ventricular Arrythmia; Cardiac Arrest With Successful Resuscitation; Sepsis; Multiple Organ Failure; Pulmonary Failure; Decompensated Heart Failure; Acute Heart Failure
Keywords: Anesthesiology; Cardiothoracic surgery; Nephrology; Perfusion; Efferentology
MeSH Terms: conditions — Shock, Cardiogenic; Sepsis; Multiple Organ Failure

STUDY DESIGN:
Intervention Model Description: Intervention team # 1 using an extracorporeal hemoperfusion device Jafron (Zhuhai Jafron Biomedical, China) (50 patients) in subgroups: A (n = 10) - patients on extracorporeal life support systems with heart failure; B (n = 10) - patients on extracorporeal life support systems with pulmonary failure; C (n = 5) - patients with implantation of a left ventricular accessory device; D (n = 25) - during operations with prolonged artificial circulation, hypothermia and circulatory arrest.
  Intervention team # 2 using extracorporeal cytokine, CytoSorb (CytoSorbents Corporation, Monmouth Junction, NJ, USA) (50 patients) in subgroups: A (n = 10) - patients on extracorporeal life support systems in heart failure; B (n = 10) - patients on extracorporeal life support systems with pulmonary failure; C (n = 5) - patients with implantation of a left ventricular accessory device; D (n = 25) - during operations with prolonged artificial circulation, hypothermia and circulatory arrest.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Intervention team (1/1 group) (Active Comparator): An extracorporeal hemoperfusion device will be installed in the device of the extracorporeal life support system for heart failure...
  (10 patients)
  Interventions: Device: HA330 - Jafron Biomedical Co., Ltd., China - extracorporeal hemocorrection
- Intervention team (1/2 group) (Active Comparator): An extracorporeal hemoperfusion device will be installed in the device of the extracorporeal life support system for pulmonary failure (10 patients).
  Interventions: Device: HA330 - Jafron Biomedical Co., Ltd., China - extracorporeal hemocorrection
- Intervention team (1/3 group) (Active Comparator): An extracorporeal hemoperfusion device will be installed in patients before/during the implantation of a left ventricular accessory (5 patients).
  Interventions: Device: HA330 - Jafron Biomedical Co., Ltd., China - extracorporeal hemocorrection
- Intervention team (1/4 group) (Active Comparator): An extracorporeal hemoperfusion device will be installed in patients during operations with prolonged artificial circulation, hypothermia, and circulatory arrest. (25 patients).
  Interventions: Device: HA330 - Jafron Biomedical Co., Ltd., China - extracorporeal hemocorrection
- Intervention team (2/1 groups) (Active Comparator): An extracorporeal hemoperfusion device will be installed in the device of the extracorporeal life support system for heart failure.
  (10 patients)
  Interventions: Device: CytoSorb (CytoSorbents Corp., USA) - an extracorporeal cytokine adsorber
- Intervention team (2/2 groups) (Active Comparator): An extracorporeal hemoperfusion device will be installed in the device of the extracorporeal life support system for pulmonary failure.
  (10 patients)
  Interventions: Device: CytoSorb (CytoSorbents Corp., USA) - an extracorporeal cytokine adsorber
- Intervention team (2/3 groups) (Active Comparator): An extracorporeal hemoperfusion device will be installed in patients before/during the implantation of a left ventricular accessory (5 patients)
  Interventions: Device: CytoSorb (CytoSorbents Corp., USA) - an extracorporeal cytokine adsorber
- Intervention team (2/4 groups) (Active Comparator): An extracorporeal hemoperfusion device will be installed in patients during operations with prolonged artificial circulation, hypothermia, and circulatory arrest. (25 patients)
  Interventions: Device: CytoSorb (CytoSorbents Corp., USA) - an extracorporeal cytokine adsorber

INTERVENTIONS:
Device: HA330 - Jafron Biomedical Co., Ltd., China - extracorporeal hemocorrection — HA330 - Jafron Biomedical Co., Ltd., China - extracorporeal hemocorrection, which is based on the removal of cytokines from whole blood by sorption on a special hemoadsorbent due to the peculiarities of its porous structure and inner surface, which is indicated in conditions where cytokine levels are extremely elevated
  Arms: Intervention team (1/1 group); Intervention team (1/2 group); Intervention team (1/3 group); Intervention team (1/4 group)
Device: CytoSorb (CytoSorbents Corp., USA) - an extracorporeal cytokine adsorber — CytoSorb (CytoSorbents Corp., USA) - an extracorporeal cytokine adsorber is a biocompatible polymer with high adsorption capacity, which is indicated in conditions where cytokine levels are extremely elevated
  Arms: Intervention team (2/1 groups); Intervention team (2/2 groups); Intervention team (2/3 groups); Intervention team (2/4 groups)

SUMMARY:
The purpose of the program. Formulation of new treatments for heart and pulmonary failure through using organ-replacing technologies.

Formulation of a clinical protocol and implementation of treatment methods into clinical practice heart and pulmonary failure using organ-replacing technologies.

New methods were created for rehabilitating the function of affected organs after implantation of the LVAD, a total artificial heart, an extracorporeal life-sustaining system will be of great importance, both for Kazakhstan and for states with similar problems of donor organ deficiency, will also improve the effectiveness of surgical treatment and reduce the level of complications and mortality of patients on the extracorporeal life-sustaining system and septic patients.

DETAILED DESCRIPTION:
Objectives of the program. Task 1. Assessment of the results of the use of extracorporeal life support systems in the treatment of pulmonary and/or heart failure.

Subtask 1.1. Assessment of the restoration of organ function during extracorporeal life support systems using extracorporeal hemocorrection.

Subtask 1.2. Assessment of the normalization of the body's immune response and restoration of organ function during extracorporeal life support systems using an extracorporeal cytokine adsorber.

Task 2. Studying the restoration of organ function during implantation of the left ventricular assist device as an organ-replacing aid in heart failure.

Subtask 2.1. Assessment of the restoration of organ function during implantation of the left ventricular assist device with the use of extracorporeal hemocorrection.

Subtask 2.2. Assessment of the normalization of the body's immune response and restoration of organ function upon implantation of the left ventricular assist device using an extracorporeal cytokine adsorber.

Task 3. Studying the restoration of organ function during the implantation of the total artificial heart as an organ-replacing aid in case of heart failure.

Task 3.1. Assessment of normalization of organ function restoration during implantation of the total artificial heart with the use of extracorporeal hemocorrection.

Task 4. Studying the restoration of organ function during operations in conditions of the long-term cardiopulmonary bypass.

Task 4.1. Assessment of the restoration of organ function during operations with long-term cardiopulmonary bypass, hypothermia, and circulatory arrest, with the use of extra corporeal hemocorrection.

Task 4.2. Assessment of the restoration of organ function during operations with long-term cardiopulmonary bypass, hypothermia, and circulatory arrest using an extracorporeal cytokine adsorber.

Task 5. Improvement of the method of implantation of organ-replacing technologies to reduce complications in the treatment of heart and pulmonary failure.

Study design. Study type: interventional (clinical study) Set of participants: 100 participants Distribution: randomized Interventional model: parallel Masking: no Primary Goal: Treatment

ELIGIBILITY:
Inclusion Criteria:

Patients on an extracorporeal life support system with heart failure:

* Implantation of intravenous ECMO
* Hemodynamic support with vasopressors and/or tonics;
* Procalcitonin level ≥ 1 ng/ml;
* Invasive hemodynamic monitoring;
* Written informed consent.

Patients on an extracorporeal life support system with pulmonary failure:

* IV ECMO implantation
* High levels of venous and arterial CO2 (CO2> 50 mmHg),
* Low paO2, SvO2, SpO2.
* Invasive hemodynamic monitoring;
* Written informed consent.

  -Patients with left ventricular assistive device implantation:
* LVAD implantation
* Biventricular heart failure IV
* INTERMACS I-III
* Hemodynamic support with vasopressors and/or tonics;
* Procalcitonin level ≥ 0.1 ng/ml;
* Invasive hemodynamic monitoring;
* Written informed consent.

  -Patients in operations with prolonged artificial circulation, hypothermia and circulatory arrest:
* Hemodynamic support with vasopressors and/or tonics;
* Bypass duration> 120 minutes
* Hypothermia ≤ 25 0С
* Circulatory arrest
* Procalcitonin level ≥ 1 ng/ml;
* Invasive hemodynamic monitoring;
* Written informed consent.

Exclusion Criteria:

* Patients on an extracorporeal life support system with heart failure:

  * Age less than 18 years old
  * Terminal hepatic or renal failure just before the procedure
  * Patient's written refusal to participate in the study
* Patients on an extracorporeal life support system with pulmonary failure:

  * Age less than 18 years old
  * Terminal hepatic or renal failure just before the procedure
  * Patient's written refusal to participate in the study
* Patients with left ventricular assistive device implantation:

  * Age less than 18 years old
  * Acute hepatic or renal failure just before the procedure
  * Patient's written refusal to participate in the study
* Patients in operations with prolonged artificial circulation, hypothermia and circulatory arrest:

  * Age less than 18 years old
  * Terminal hepatic or renal failure just before the procedure
  * Patient's written refusal to participate in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-07-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Extracorporeal life support system with pulmonary and / or heart failure: Cytokine response | 24-48 hours
  The level of pro- and anti-inflammatory cytokines (IL-1, IL-6, IL-8, IL-10, tumor alpha-factor) before the start, 2 hours after the start of ECMO support, when ECMO is turned off, 24 hours after ECMO is turned off.
Extracorporeal life support system with pulmonary and / or heart failure: SOFA-Score | 24, 48, 72 hours
  Sequential Organ Failure Assessment Score at 24, 48, 72 h (values from 6 to 24, where the higher values explain higher disease severity)
Extracorporeal life support system with pulmonary and / or heart failure | Time: first 72 hours
  Doses of vasopressors and / or inotropes (µg / h / kg bodyweight)
Patients with left ventricular assist device implantation: Difference of Cytokine response | 24-48 hours
  Level of pro- and anti-inflammatory cytokines (IL-1, IL-6, IL-8, IL-10, tumor necrosis factor-alfa, procalcitonin)
Patients with left ventricular assist device implantation:vasopressors and / or inotropes | first 72 hours
  Doses of vasopressors and / or inotropes (µg / h / kg bodyweight)
Patients with left ventricular assist device implantation:Renal function | first 72 hours
  creatinine level
Patients with left ventricular assist device implantation:Lactate level | first 72 hours
  Lactate level
For operations with prolonged artificial circulation, hypothermia and circulatory arrest: Difference of Cytokine response | 24-48 hours
  Level of pro- and anti-inflammatory cytokines (IL-1, IL-6, IL-8, IL-10, tumor necrosis factor-alfa, procalcitonin, C-reactive protein)
For operations with prolonged artificial circulation, hypothermia and circulatory arrest: SOFA-Score | 24, 48, 72 hours
  Sequential Organ Failure Assessment Score at 24, 48, 72 h (values from 6 to 24, where the higher values explain higher disease severity)
Extracorporeal life support system with pulmonary and / or heart failure:Difference of mean arterial pressure | 24, 48, 72 hours
  Comparison of mean arterial pressure at 24, 48, 72 hours between between two interventions (CytoSorb and Jafron)
Extracorporeal life support system with pulmonary and / or heart failure: Difference of CVP | 24, 48, 72 hours
  Comparison of CVP at 24, 48, 72 hours between between two interventions (CytoSorb and Jafron)
Extracorporeal life support system with pulmonary and / or heart failure: Serum lactate | 24, 48, 72 hours
  Level of serum lactate at 24, 48, 72 h
Extracorporeal life support system with pulmonary and / or heart failure:Days on ventilator, vasopressor and renal replacement therapy | until day 30 post-surgery
  Total days on ventilator, vasopressor and renal replacement therapy within 30 days post-surgery will be assessed
For operations with prolonged artificial circulation, hypothermia and circulatory arrest: Difference of mean arterial pressure | 24, 48, 72 hours
  Comparison of mean arterial pressure at 24, 48, 72 hours between between two interventions (CytoSorb and Jafron)
For operations with prolonged artificial circulation, hypothermia and circulatory arrest: Difference of CVP | 24, 48, 72 hours
  Comparison of mean arterial pressure at 24, 48, 72 hours between between two interventions (CytoSorb and Jafron)
For operations with prolonged artificial circulation, hypothermia and circulatory arrest: Level of Serum lactate | 24, 48, 72 hours
  Comparison of mean arterial pressure at 24, 48, 72 hours between between two interventions (CytoSorb and Jafron)

SECONDARY OUTCOMES:
Extracorporeal life support system with pulmonary and / or heart failure:The level of C-reactive protein (CRP) | 24-48 hours
  The level of C-reactive protein (CRP) before the start of ECMO, 2 hours after the implantation of ECMO, during ECMO, 24 hours after ECMO explantation.
Extracorporeal life support system with pulmonary and / or heart failure: Level of leukocyte | 24-48 hours
  Level of leukocyte cells in the bloodstream at 24, 48 hours
Extracorporeal life support system with pulmonary and / or heart failure:Application and dosage of vasopressors | first 48 hours
  Incidence of application and level of dosage of vasopressors on days 2 and 3 after surgery
Patients with left ventricular assist device implantation: The level of C-reactive protein (CRP) | 24-48 hours
  The level of C-reactive protein (CRP) before the start of the operation, 2 hours after the start of the operation, when the operation is turned off, 24 hours after the shutdown of the operation
Patients with left ventricular assist device implantation: Application and dosage of vasopressors | first 48 hours
  Incidence of application and level of dosage of vasopressors on days 2 and 3 after surgery
For operations with prolonged artificial circulation, hypothermia and circulatory arrest: The level of C-reactive protein (CRP) | 24-48 hours
  The level of C-reactive protein (CRP) before the cardiopulmonary bypass 2 hours after the cardiopulmonary bypass, when the cardiopulmonary bypass is turned off, 24 hours after the cardiopulmonary bypass.
For operations with prolonged artificial circulation, hypothermia and circulatory arrest:Leukocyte function | first 48 hours
  Leukocyte function: heterogeneity of the population of leukocyte cells in the bloodstream
For operations with prolonged artificial circulation, hypothermia and circulatory arrest: Application and dosage of vasopressors | first 48 hours
  Incidence of application and level of dosage of vasopressors on days 2 and 3 after surgery
Extracorporeal life support system with pulmonary and / or heart failure:The level of leukocytes | 24-48 hours
  The level of leukocytes before the start of ECMO, 2 hours after the implantation of ECMO, during ECMO, 24 hours after ECMO explantation
Extracorporeal life support system with pulmonary and / or heart failure:The level of procalcitonin | 24-48 hours
  The level of procalcitonin before the start of ECMO, 2 hours after the implantation of ECMO, during ECMO, 24 hours after ECMO explantation.
Extracorporeal life support system with pulmonary and / or heart failure:Application and dosage of inotropes | first 48 hours
  Incidence of application and level of dosage of inotropes on days 2 and 3 after surgery
Patients with left ventricular assist device implantation: The level of leukocytes | 24-48 hours
  The level of leukocytes before the start of the operation, 2 hours after the start of the operation, when the operation is turned off, 24 hours after the shutdown of the operation
Patients with left ventricular assist device implantation: The level of procalcitonin | 24-48 hours
  The level of procalcitonin before the start of the operation, 2 hours after the start of the operation, when the operation is turned off, 24 hours after the shutdown of the operation
Patients with left ventricular assist device implantation: Application and dosage of inotropes | first 48 hours
  Incidence of application and level of dosage of inotropes on days 2 and 3 after surgery
For operations with prolonged cardio pulmonary bypass, hypothermia and circulatory arrest: The level of leukocytes | 24-48 hours
  The level of leukocytes before the cardiopulmonary bypass 2 hours after the cardiopulmonary bypass, when the cardiopulmonary bypass is turned off, 24 hours after the cardiopulmonary bypass.
For operations with prolonged cardiopulmonary bypass, hypothermia, and circulatory arrest: The level of procalcitonin | 24-48 hours
  The level of procalcitonin before the cardiopulmonary bypass 2 hours after the cardiopulmonary bypass, when the cardiopulmonary bypass is turned off, 24 hours after the cardiopulmonary bypass.
For operations with prolonged cardiopulmonary bypass, hypothermia, and circulatory arrest: Application and dosage of inotropes | first 48 hours
  Incidence of application and level of dosage of inotropes on days 2 and 3 after surgery

OTHER OUTCOMES:
Length of stay | first 48 hours
  Length of stay in the intensive care unit
Length of hospital stay | up to 1 month
  Length of hospital stay
30 day survival rate. | 30 day
  30 day survival rate.

CONTACTS AND LOCATIONS:
Overall Officials: Yuri Pya, PhD, MD, Principal Investigator — National research Center for Cardiac Surgery JSC
Locations (1):
- National Research Center For Cardiac Surgery, Astana, Kazakhstan

IPD SHARING:
Plan to Share IPD: Yes
Yes: There is a plan to make IPD and related data dictionaries available.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: from October 2021 year and will become available till December 2023 year.
Access Criteria: The resulting patient data will be strictly confidential with ensuring privacy through strictly limited access to data, de-identification of data and destruction after the end of the study.
URL: http://heartcenter.kz

REFERENCES:
- [Result] Starling RC. Improved quantity and quality of life: a winning combination to treat advanced heart failure. J Am Coll Cardiol. 2010 Apr 27;55(17):1835-6. doi: 10.1016/j.jacc.2010.03.010. No abstract available. PMID 20413034
- [Result] Maciver J, Ross HJ. Quality of life and left ventricular assist device support. Circulation. 2012 Aug 14;126(7):866-74. doi: 10.1161/CIRCULATIONAHA.111.040279. No abstract available. PMID 22891167
- [Result] Tozzi P, Hullin R. Mechanical circulatory support for destination therapy. Swiss Med Wkly. 2016 Mar 5;146:w14267. doi: 10.4414/smw.2016.14267. eCollection 2016. PMID 26945160
- [Result] Paolone S. Extracorporeal Membrane Oxygenation (ECMO) for Lung Injury in Severe Acute Respiratory Distress Syndrome (ARDS): Review of the Literature. Clin Nurs Res. 2017 Dec;26(6):747-762. doi: 10.1177/1054773816677808. Epub 2016 Nov 11. PMID 27836935
- [Result] Abrams D, Garan AR, Abdelbary A, Bacchetta M, Bartlett RH, Beck J, Belohlavek J, Chen YS, Fan E, Ferguson ND, Fowles JA, Fraser J, Gong M, Hassan IF, Hodgson C, Hou X, Hryniewicz K, Ichiba S, Jakobleff WA, Lorusso R, MacLaren G, McGuinness S, Mueller T, Park PK, Peek G, Pellegrino V, Price S, Rosenzweig EB, Sakamoto T, Salazar L, Schmidt M, Slutsky AS, Spaulding C, Takayama H, Takeda K, Vuylsteke A, Combes A, Brodie D; International ECMO Network (ECMONet) and The Extracorporeal Life Support Organization (ELSO). Position paper for the organization of ECMO programs for cardiac failure in adults. Intensive Care Med. 2018 Jun;44(6):717-729. doi: 10.1007/s00134-018-5064-5. Epub 2018 Feb 15. PMID 29450594
- [Result] Hunt SA. Taking heart--cardiac transplantation past, present, and future. N Engl J Med. 2006 Jul 20;355(3):231-5. doi: 10.1056/NEJMp068048. No abstract available. PMID 16855261
- [Result] Hunt SA, Haddad F. The changing face of heart transplantation. J Am Coll Cardiol. 2008 Aug 19;52(8):587-98. doi: 10.1016/j.jacc.2008.05.020. PMID 18702960
- [Result] Lund LH, Edwards LB, Kucheryavaya AY, Benden C, Christie JD, Dipchand AI, Dobbels F, Goldfarb SB, Levvey BJ, Meiser B, Yusen RD, Stehlik J; International Society of Heart and Lung Transplantation. The registry of the International Society for Heart and Lung Transplantation: thirty-first official adult heart transplant report--2014; focus theme: retransplantation. J Heart Lung Transplant. 2014 Oct;33(10):996-1008. doi: 10.1016/j.healun.2014.08.003. Epub 2014 Aug 14. No abstract available. PMID 25242124
- [Result] Sogayar AM, Machado FR, Rea-Neto A, Dornas A, Grion CM, Lobo SM, Tura BR, Silva CL, Cal RG, Beer I, Michels V, Safi J, Kayath M, Silva E; Costs Study Group - Latin American Sepsis Institute. A multicentre, prospective study to evaluate costs of septic patients in Brazilian intensive care units. Pharmacoeconomics. 2008;26(5):425-34. doi: 10.2165/00019053-200826050-00006. PMID 18429658
- [Result] Khwannimit B, Bhurayanontachai R. The direct costs of intensive care management and risk factors for financial burden of patients with severe sepsis and septic shock. J Crit Care. 2015 Oct;30(5):929-34. doi: 10.1016/j.jcrc.2015.05.011. Epub 2015 May 20. PMID 26051981
- [Result] Iskander KN, Osuchowski MF, Stearns-Kurosawa DJ, Kurosawa S, Stepien D, Valentine C, Remick DG. Sepsis: multiple abnormalities, heterogeneous responses, and evolving understanding. Physiol Rev. 2013 Jul;93(3):1247-88. doi: 10.1152/physrev.00037.2012. PMID 23899564
- [Result] Kwan A, Hubank M, Rashid A, Klein N, Peters MJ. Transcriptional instability during evolving sepsis may limit biomarker based risk stratification. PLoS One. 2013;8(3):e60501. doi: 10.1371/journal.pone.0060501. Epub 2013 Mar 27. PMID 23544148
- [Result] Akira S, Uematsu S, Takeuchi O. Pathogen recognition and innate immunity. Cell. 2006 Feb 24;124(4):783-801. doi: 10.1016/j.cell.2006.02.015. PMID 16497588
- [Result] Hotchkiss RS, Monneret G, Payen D. Sepsis-induced immunosuppression: from cellular dysfunctions to immunotherapy. Nat Rev Immunol. 2013 Dec;13(12):862-74. doi: 10.1038/nri3552. Epub 2013 Nov 15. PMID 24232462
- [Result] Venet F, Lukaszewicz AC, Payen D, Hotchkiss R, Monneret G. Monitoring the immune response in sepsis: a rational approach to administration of immunoadjuvant therapies. Curr Opin Immunol. 2013 Aug;25(4):477-83. doi: 10.1016/j.coi.2013.05.006. Epub 2013 May 28. PMID 23725873
- [Result] Laszlo I, Trasy D, Molnar Z, Fazakas J. Sepsis: From Pathophysiology to Individualized Patient Care. J Immunol Res. 2015;2015:510436. doi: 10.1155/2015/510436. Epub 2015 Jul 15. PMID 26258150
- [Result] Cruz DN, Antonelli M, Fumagalli R, Foltran F, Brienza N, Donati A, Malcangi V, Petrini F, Volta G, Bobbio Pallavicini FM, Rottoli F, Giunta F, Ronco C. Early use of polymyxin B hemoperfusion in abdominal septic shock: the EUPHAS randomized controlled trial. JAMA. 2009 Jun 17;301(23):2445-52. doi: 10.1001/jama.2009.856. PMID 19531784
- [Result] Bellomo R, Baldwin I, Ronco C. Extracorporeal blood purification therapy for sepsis and systemic inflammation: its biological rationale. Contrib Nephrol. 2001;(132):367-74. doi: 10.1159/000060105. PMID 11395904
- [Result] Namas RA, Namas R, Lagoa C, Barclay D, Mi Q, Zamora R, Peng Z, Wen X, Fedorchak MV, Valenti IE, Federspiel WJ, Kellum JA, Vodovotz Y. Hemoadsorption reprograms inflammation in experimental gram-negative septic peritonitis: insights from in vivo and in silico studies. Mol Med. 2012 Dec 20;18(1):1366-74. doi: 10.2119/molmed.2012.00106. PMID 22751621
- [Result] Peng ZY, Carter MJ, Kellum JA. Effects of hemoadsorption on cytokine removal and short-term survival in septic rats. Crit Care Med. 2008 May;36(5):1573-7. doi: 10.1097/CCM.0b013e318170b9a7. PMID 18434884
- [Result] Peng ZY, Wang HZ, Carter MJ, Dileo MV, Bishop JV, Zhou FH, Wen XY, Rimmele T, Singbartl K, Federspiel WJ, Clermont G, Kellum JA. Acute removal of common sepsis mediators does not explain the effects of extracorporeal blood purification in experimental sepsis. Kidney Int. 2012 Feb;81(4):363-9. doi: 10.1038/ki.2011.320. Epub 2011 Sep 14. PMID 21918497
- [Result] Kellum JA, Venkataraman R, Powner D, Elder M, Hergenroeder G, Carter M. Feasibility study of cytokine removal by hemoadsorption in brain-dead humans. Crit Care Med. 2008 Jan;36(1):268-72. doi: 10.1097/01.CCM.0000291646.34815.BB. PMID 18090355
- [Result] Friesecke S, Trager K, Schittek GA, Molnar Z, Bach F, Kogelmann K, Bogdanski R, Weyland A, Nierhaus A, Nestler F, Olboeter D, Tomescu D, Jacob D, Haake H, Grigoryev E, Nitsch M, Baumann A, Quintel M, Schott M, Kielstein JT, Meier-Hellmann A, Born F, Schumacher U, Singer M, Kellum J, Brunkhorst FM. International registry on the use of the CytoSorb(R) adsorber in ICU patients : Study protocol and preliminary results. Med Klin Intensivmed Notfmed. 2019 Nov;114(8):699-707. doi: 10.1007/s00063-017-0342-5. Epub 2017 Sep 4. PMID 28871441
- [Result] Rhodes A, Evans LE, Alhazzani W, Levy MM, Antonelli M, Ferrer R, Kumar A, Sevransky JE, Sprung CL, Nunnally ME, Rochwerg B, Rubenfeld GD, Angus DC, Annane D, Beale RJ, Bellinghan GJ, Bernard GR, Chiche JD, Coopersmith C, De Backer DP, French CJ, Fujishima S, Gerlach H, Hidalgo JL, Hollenberg SM, Jones AE, Karnad DR, Kleinpell RM, Koh Y, Lisboa TC, Machado FR, Marini JJ, Marshall JC, Mazuski JE, McIntyre LA, McLean AS, Mehta S, Moreno RP, Myburgh J, Navalesi P, Nishida O, Osborn TM, Perner A, Plunkett CM, Ranieri M, Schorr CA, Seckel MA, Seymour CW, Shieh L, Shukri KA, Simpson SQ, Singer M, Thompson BT, Townsend SR, Van der Poll T, Vincent JL, Wiersinga WJ, Zimmerman JL, Dellinger RP. Surviving Sepsis Campaign: International Guidelines for Management of Sepsis and Septic Shock: 2016. Intensive Care Med. 2017 Mar;43(3):304-377. doi: 10.1007/s00134-017-4683-6. Epub 2017 Jan 18. PMID 28101605
- [Result] Moreno R, Vincent JL, Matos R, Mendonca A, Cantraine F, Thijs L, Takala J, Sprung C, Antonelli M, Bruining H, Willatts S. The use of maximum SOFA score to quantify organ dysfunction/failure in intensive care. Results of a prospective, multicentre study. Working Group on Sepsis related Problems of the ESICM. Intensive Care Med. 1999 Jul;25(7):686-96. doi: 10.1007/s001340050931. PMID 10470572
- [Result] Hetz H, Berger R, Recknagel P, Steltzer H. Septic shock secondary to beta-hemolytic streptococcus-induced necrotizing fasciitis treated with a novel cytokine adsorption therapy. Int J Artif Organs. 2014 May;37(5):422-6. doi: 10.5301/ijao.5000315. Epub 2014 Apr 17. PMID 24811308
- [Result] Kogelmann K, Jarczak D, Scheller M, Druner M. Hemoadsorption by CytoSorb in septic patients: a case series. Crit Care. 2017 Mar 27;21(1):74. doi: 10.1186/s13054-017-1662-9. PMID 28343448
- [Result] David S, Thamm K, Schmidt BMW, Falk CS, Kielstein JT. Effect of extracorporeal cytokine removal on vascular barrier function in a septic shock patient. J Intensive Care. 2017 Jan 21;5:12. doi: 10.1186/s40560-017-0208-1. eCollection 2017. PMID 28127437
- [Result] Nemeth E, Kovacs E, Racz K, Soltesz A, Szigeti S, Kiss N, Csikos G, Koritsanszky KB, Berzsenyi V, Trembickij G, Fabry S, Prohaszka Z, Merkely B, Gal J. Impact of intraoperative cytokine adsorption on outcome of patients undergoing orthotopic heart transplantation-an observational study. Clin Transplant. 2018 Apr;32(4):e13211. doi: 10.1111/ctr.13211. Epub 2018 Feb 27. PMID 29377282
- [Result] Trasy D, Tanczos K, Nemeth M, Hankovszky P, Lovas A, Mikor A, Laszlo I, Hajdu E, Osztroluczki A, Fazakas J, Molnar Z; EProK study group. Early procalcitonin kinetics and appropriateness of empirical antimicrobial therapy in critically ill patients: A prospective observational study. J Crit Care. 2016 Aug;34:50-5. doi: 10.1016/j.jcrc.2016.04.007. Epub 2016 Apr 13. PMID 27288610
- [Result] Riedel S. Procalcitonin and the role of biomarkers in the diagnosis and management of sepsis. Diagn Microbiol Infect Dis. 2012 Jul;73(3):221-7. doi: 10.1016/j.diagmicrobio.2012.05.002. PMID 22704255
- [Result] Nylen ES, Whang KT, Snider RH Jr, Steinwald PM, White JC, Becker KL. Mortality is increased by procalcitonin and decreased by an antiserum reactive to procalcitonin in experimental sepsis. Crit Care Med. 1998 Jun;26(6):1001-6. doi: 10.1097/00003246-199806000-00015. PMID 9635646
- [Result] Schadler D, Pausch C, Heise D, Meier-Hellmann A, Brederlau J, Weiler N, Marx G, Putensen C, Spies C, Jorres A, Quintel M, Engel C, Kellum JA, Kuhlmann MK. The effect of a novel extracorporeal cytokine hemoadsorption device on IL-6 elimination in septic patients: A randomized controlled trial. PLoS One. 2017 Oct 30;12(10):e0187015. doi: 10.1371/journal.pone.0187015. eCollection 2017. PMID 29084247
- [Result] Trasy D, Molnar Z. Procalcitonin - Assisted Antibiotic Strategy in Sepsis. EJIFCC. 2017 May 1;28(2):104-113. eCollection 2017 May. PMID 28757818
- [Result] Tschaikowsky K, Sagner S, Lehnert N, Kaul M, Ritter J. Endothelin in septic patients: effects on cardiovascular and renal function and its relationship to proinflammatory cytokines. Crit Care Med. 2000 Jun;28(6):1854-60. doi: 10.1097/00003246-200006000-00028. PMID 10890632
- [Result] Benjamin EJ, Virani SS, Callaway CW, Chamberlain AM, Chang AR, Cheng S, Chiuve SE, Cushman M, Delling FN, Deo R, de Ferranti SD, Ferguson JF, Fornage M, Gillespie C, Isasi CR, Jimenez MC, Jordan LC, Judd SE, Lackland D, Lichtman JH, Lisabeth L, Liu S, Longenecker CT, Lutsey PL, Mackey JS, Matchar DB, Matsushita K, Mussolino ME, Nasir K, O'Flaherty M, Palaniappan LP, Pandey A, Pandey DK, Reeves MJ, Ritchey MD, Rodriguez CJ, Roth GA, Rosamond WD, Sampson UKA, Satou GM, Shah SH, Spartano NL, Tirschwell DL, Tsao CW, Voeks JH, Willey JZ, Wilkins JT, Wu JH, Alger HM, Wong SS, Muntner P; American Heart Association Council on Epidemiology and Prevention Statistics Committee and Stroke Statistics Subcommittee. Heart Disease and Stroke Statistics-2018 Update: A Report From the American Heart Association. Circulation. 2018 Mar 20;137(12):e67-e492. doi: 10.1161/CIR.0000000000000558. Epub 2018 Jan 31. No abstract available. PMID 29386200
- [Result] Rodriguez LE, Suarez EE, Loebe M, Bruckner BA. Ventricular assist devices (VAD) therapy: new technology, new hope? Methodist Debakey Cardiovasc J. 2013 Jan-Mar;9(1):32-7. doi: 10.14797/mdcj-9-1-32. PMID 23519193
- [Result] Lietz K, Long JW, Kfoury AG, Slaughter MS, Silver MA, Milano CA, Rogers JG, Naka Y, Mancini D, Miller LW. Outcomes of left ventricular assist device implantation as destination therapy in the post-REMATCH era: implications for patient selection. Circulation. 2007 Jul 31;116(5):497-505. doi: 10.1161/CIRCULATIONAHA.107.691972. Epub 2007 Jul 16. PMID 17638928
- [Result] Feldman D, Pamboukian SV, Teuteberg JJ, Birks E, Lietz K, Moore SA, Morgan JA, Arabia F, Bauman ME, Buchholz HW, Deng M, Dickstein ML, El-Banayosy A, Elliot T, Goldstein DJ, Grady KL, Jones K, Hryniewicz K, John R, Kaan A, Kusne S, Loebe M, Massicotte MP, Moazami N, Mohacsi P, Mooney M, Nelson T, Pagani F, Perry W, Potapov EV, Eduardo Rame J, Russell SD, Sorensen EN, Sun B, Strueber M, Mangi AA, Petty MG, Rogers J; International Society for Heart and Lung Transplantation. The 2013 International Society for Heart and Lung Transplantation Guidelines for mechanical circulatory support: executive summary. J Heart Lung Transplant. 2013 Feb;32(2):157-87. doi: 10.1016/j.healun.2012.09.013. No abstract available. PMID 23352391
- [Result] Hetzer R, Delmo Walter EM. Trends and outcomes in heart transplantation: the Berlin experience. HSR Proc Intensive Care Cardiovasc Anesth. 2013;5(2):76-80. PMID 23888228
- [Result] Chen YF, Tsai WC, Lin CC, Tsai LY, Lee CS, Huang CH, Pan PC, Chen ML. Effect of leukocyte depletion on endothelial cell activation and transendothelial migration of leukocytes during cardiopulmonary bypass. Ann Thorac Surg. 2004 Aug;78(2):634-42; discussion 642-3. doi: 10.1016/j.athoracsur.2004.02.091. PMID 15276536

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-01-01): https://cdn.clinicaltrials.gov/large-docs/30/NCT05090930/Prot_SAP_000.pdf
  • Informed Consent Form (2021-01-01): https://cdn.clinicaltrials.gov/large-docs/30/NCT05090930/ICF_001.pdf